CLINICAL TRIAL: NCT04138303
Title: The Effects of a Calorie-Restrictive Low-Carbohydrate Diet Versus an Unrestrictive Ancestral Diet on Microbiota and Cardiometabolic Disease Markers of Obese Individuals Performing an Intense Exercise Program
Brief Title: Exercise and Nutrition on Obese Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Wesley Smith, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20190936
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Only Group (EX) (Experimental): Participants will only receive the exercise protocol without nutrition education or counseling and instructed to continue to consume their regular diet.
  Interventions: Other: Exercise Protocol
- Exercise with CR-LC Group (Experimental): Participants will receive the exercise protocol and CR-LC Diet regimen.
  Interventions: Other: Exercise Protocol; Other: Calorie-Restrictive Low Carbohydrate Diet (CR-LC)
- Exercise with Ancestral Diet (AD) Group (Experimental): Participants will receive the exercise protocol and AD regimen.
  Interventions: Other: Exercise Protocol; Other: Ancestral Diet (AD)

INTERVENTIONS:
Other: Exercise Protocol — The exercise protocol consists of a nine-week progressive intense-conditioning program involving six consecutive days (Monday-Saturday) of one-hour exercises and one-day rest weekly for a total of 54 days of exercise. Exercises are performed in person as a group with other participating subjects and lead by certified instructors. Exercises will involve a variety of activities ranging from running, cycling, whole-body functional movements, power movements, and open-chain weight lifting with barbells and resistance bands.
Other: Calorie-Restrictive Low Carbohydrate Diet (CR-LC) — Consists of weekly nutrition plans, counseling and monitoring by on-site registered dietitians and nutritionists for nine weeks. CR-LC consists of caloric and macronutrient restrictions. Caloric restrictions involves a 40% deficit from calculated total daily energy expenditure. Macronutrient restriction involves a high protein, low carbohydrate diet (35% protein, 25% carbohydrate and 40% fat).
  Arms: Exercise with CR-LC Group
Other: Ancestral Diet (AD) — Consists of weekly nutrition plans, counseling and monitoring by on-site registered dietitians and nutritionists for nine weeks. AD consists of consuming only whole foods and avoiding processed foods. Emphasis will be on food quality with no caloric or macronutrient restrictions.
  Arms: Exercise with Ancestral Diet (AD) Group

SUMMARY:
The purpose of this study is to examine the effects nine weeks of intense exercise training will have on weight, inflammation, and intestinal bacteria composition of overweight and obese adults.

ELIGIBILITY:
Inclusion criteria:

1. Individuals who are overweight (BMI ≥ 25) and/or obese (BMI ≥ 30).
2. Individuals who volunteer for the 54-day exercise program.
3. Individuals with no history of diabetes mellitus (type I or II) or sickle cell disease.
4. Individuals who are not taking antibiotics and have not taken antibiotics within 3 months.
5. Individuals who are not taking probiotics.
6. Individuals who are not taking Metformin.
7. Individuals who are cleared by their physician to perform strenuous exercise.
8. Individuals with no physically debilitating injuries that would keep them from being able to perform the exercises prescribed.
9. Individuals who are between 18 and 60.

Exclusion criteria:

1. Any subjects who do not meet all of the inclusion criteria and/or are unable to consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

PRIMARY OUTCOMES:
Change in fecal microbiota diversity | Baseline, 9 weeks
  Change in fecal microbiota alpha-diversity will be assessed via stool sample evaluation
Change in Bacteriodetes/Firmicutes ratio | Baseline, 9 weeks
  Change in Bacteriodetes/Firmicutes ratio as assessed via stool sample evaluation
Percent change in fecal microbiota composition | Baseline, 9 weeks
  Percent change in Bacteriodetes phyla and percent change of short-chain fatty acid-producing species as assessed via stool sample evaluation
Change in inflammatory markers | Baseline, 9 weeks
  Change in serum inflammatory markers including Interleukin (IL)-1ß, IL-6, Tumor Necrosis Factor (TNF)-α and liposaccharide (LPS) evaluated in pg/ml.
Change in leptin/adiponectin ratio | Baseline, 9 weeks
  Change in serum adipose markers assessed as change in leptin/adiponectin ratio.
Correlation of serum triglycerides with leptin levels | Baseline, 9 weeks
  The correlation of the serum triglyceride levels will be evaluated against serum leptin levels.
Change in body weight | Baseline, 9 weeks
  Change in body composition as evaluated as change in body weight measured in lbs.
Change in resting metabolic rate | Baseline, 9 weeks
  Change in body composition as evaluated as change in resting metabolic rate measured in Calories per day.
Change in body composition | Baseline, 9 weeks
  Change in body composition as evaluated as change in body fat and lean body mass percentage
Change in waist circumference | Baseline, 9 weeks
  Change in waist circumference measured in inches.
Change in blood pressure | Baseline, 9 weeks
  Change in blood pressure assessed as systolic and diastolic pressure in mmHg.
Change in visceral fat | Baseline, 9 weeks
  Change in visceral fat levels will be measured using InBody570 with scores ranging from 1-20, with the higher score indicating increased visceral fat (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Smith, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No